CLINICAL TRIAL: NCT04962685
Title: Evaluation of Masticatory Muscle Activity in Patients With Unilateral Posterior Crossbite Before and After Rapid Maxillary Expansion
Brief Title: Evaluation of Muscle Activity in Unilateral Posterior Crossbite
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Albert Pérez Bellmunt, Principal Investigator, Universitat Internacional de Catalunya
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CER202108
Record Dates: First submitted 2021-06-22; First posted 2021-07-15 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Malocclusion; Muscle Activity; Maxillary Expansion
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unilateral Posterior Crossbite (Experimental)
  Interventions: Other: Rapid Maxillary Expansion
- Normal occlusion (No Intervention)

INTERVENTIONS:
Other: Rapid Maxillary Expansion — Subjects in the experimental group (with unilateral posterior crossbite) will be treated with Maxillary Rapid Expansion using a disjunctor fixed with two bands on the upper first permanent molars and a mesh cemented to the upper first premolars or upper first primary molars (depending on the eruptive stage of the patient).
  The breaker screw will be activated twice a day until a transverse overcorrection of 2 mm is achieved in the first permanent molars. When the active disjunction phase is completed, the screw will be blocked out with light-curing flowable resin and the patient will wear the cemented disjunctor as a retainer for a minimum of six months.
  Arms: Unilateral Posterior Crossbite

SUMMARY:
Posterior crossbite (PCB) is defined as the presence of one or more teeth of the posterior group (canine to third molar) in an inverted buccolingual relationship, where the vestibular cusp of the upper tooth is in contact with the central fossa of its lower antagonist tooth. It is one of the most common malocclusions in children, with a prevalence of 8 to 22% among orthodontic patients in primary and mixed dentition and 5 to 15% among the general population. It can be bilateral (MCPB) or unilateral (MCPU). In 71-84% of cases, CCM in growing patients appears as a functional CCBM and is therefore associated with a functional mandibular deviation.

The hypothesis of this study is, that unilateral posterior crossbite correction by Rapid Maxillary expansion achieves improved symmetry and muscle activation potential in treated patients.

The objective of this study is to evaluate the muscle activity of masticatory muscles in patients with unilateral posterior crossbite with superficial electromyography before and after treatment with rapid maxillary expansion.

Superficial electromyography will be measured in masseter and temporalis muscle before treatment, when the patients bite is corrected and after the treatment.

Three static and two dynamic tasks will be measured.

DETAILED DESCRIPTION:
Posterior crossbite (PCB) is defined as the presence of one or more teeth of the posterior group (canine to third molar) in an inverted buccolingual relationship, where the vestibular cusp of the upper tooth is in contact with the central fossa of its lower antagonist tooth. It is one of the most common malocclusions in children, with a prevalence of 8 to 22% among orthodontic patients in primary and mixed dentition and 5 to 15% among the general population. It can be bilateral (MCPB) or unilateral (MCPU). In 71-84% of cases, CCM in growing patients appears as a functional CCBM, and is therefore associated with a functional mandibular deviation.

There is evidence that an altered relationship between upper and lower teeth is associated with differences in the temporomandibular condyle-temporomandibular fossa relationship between the right and left sides. Asymmetric masticatory function in patients with CCM has been related to differences in development between the right and left sides of the mandibular bone during growth, asymmetric contraction of the masticatory musculature, decreased thickness of the cross-sided masseter muscle and altered masticatory pattern. Therefore, previous studies suggest that UCPM may contribute to the development of skeletal asymmetries and temporomandibular disorders (TMD). Given that the most frequent cause of UCPD is the reduction in maxillary width, other authors conclude that early treatment with Rapid Maxillary Expansion (RME) would be recommended to reduce the risk of developing TMD and craniofacial anomalies in adulthood, due to postural alterations and asymmetric function and growth of skeletal and muscular structures.

Muscle activity is commonly recorded in research using surface electromyography (sEMG). sEMG has previously been used in similar studies because it is less invasive than intramuscular electromyography. However, sEMG data can be affected by various artifacts, resulting in questionable interpretation of the results. For this reason, Ferrario et al. described a method to standardize myoelectric potentials, with indices that record the activation of the levator muscles and the level of symmetry in activation between contralateral muscle pairs. This protocol reduces within-sample variability and can be used for the assessment of masticatory muscle activity during static and dynamic tasks.

The hypotheses of this study are:

Patients with unilateral posterior crossbite have less activity of masseter and anterior temporalis muscles during masticatory function than patients with normal occlusion.

Patients with unilateral posterior crossbite have a greater asymmetry in the masticatory function of masseter and anterior temporalis muscles than patients with normal occlusion.

The correction of unilateral posterior crossbite by Rapid Maxillary Expansion achieves an improvement in the symmetry and muscle activation potential of the treated patients.

The masticatory muscle function of patients treated with ERM offers values comparable to those of patients with normal occlusion.

The main objectives of this study are:

To evaluate the activity of the masseter and anterior temporalis muscles of infant patients with unilateral posterior crossbite, before and after correction with Rapid Maxillary Expansion, using surface electromyography and a standardized protocol.

To evaluate whether the presence of unilateral posterior crossbite is associated with less symmetrical activation of the masseter and anterior temporalis muscles, comparing the activity of these muscles in patients with unilateral posterior crossbite with a control group with normal occlusion.

To evaluate whether unilateral posterior crossbite correction can improve the function of the masseter and anterior temporalis muscles by comparing the patient to himself/herself pre- and post-correction of the unilateral posterior crossbite with Rapid Maxillary Expansion.

To evaluate whether the patient who has undergone Maxillary Rapid Expansion has masseter and anterior temporalis muscle function comparable to that of patients with normal occlusion, comparing patients treated with ERM to control patients with normal occlusion.

Dental exam:

In the experimental group, posterior crossbite will be diagnosed clinically by the presence of at least one posterior tooth in complete crossbite, with the vestibular cusp of the upper tooth occluding lingually from the vestibular cusp of the lower antagonist tooth.

Mandibular laterodeviation will be diagnosed by the Dawson maneuver. This clinical maneuver is commonly used to distinguish between functional or morphological crossbite and to detect centric relation (CR) position and the discrepancy between CR and maximum intercuspidation position (MIP). In the present study, since the investigators want to evaluate the effect of crossbite with mandibular laterodeviation on masticatory muscle activity, the subjects in the experimental group will present a functional mandibular deviation between CR and MIP, with a complete unilateral posterior crossbite in MIP, but incomplete in CR.

Electromyography will be performed using the mDurance® surface electromyograph (mDurance Solutions SL; Granada, Spain) in order to capture muscle activity of the superficial masseter muscle (M) and the anterior temporalis muscle (AT) bilaterally and simultaneously during standardized tasks.

Bipolar surface electrodes prepared with Ag/AgCl gel will be used. In order to reduce the impedance of the electrodes, the patient's skin will be carefully cleaned with a cotton swab soaked in alcohol before electrode placement. The tests will be performed at least five minutes later, to allow the conductive gel to prepare the skin surface adequately. The electrodes will have a diameter of 10 mm and an interelectrode distance of 20 ± 1 mm. They will be positioned on the muscle bellies according to the protocol described by Ferrario et al. as follows:

Masseter muscle: the operator, standing behind the seated subject, will palpate the muscle belly while the subject clenches his teeth. He will then fix the electrode, parallel to the muscle fibers, about 3 cm superiorly and anteriorly to the mandibular angle, with the upper pole of the electrode at the intersection between the tragus-labial commissure and exocantion-gonion lines.

Anterior temporalis muscle: the operator, standing behind the seated subject, will palpate the muscle belly while the subject clenches the teeth. The electrode will be fixed vertically along the anterior margin of the muscle (corresponding to the frontoparietal suture).

The ground electrode will be positioned on the forehead. This position has been shown to be optimal for electrode configuration and the protocol of Ferrario et al. has been used in many similar studies, allowing useful comparisons between different subjects and studies.

The sEMG protocol will include three static and two dynamic tests.

The static tests will be as follows:

Resting activity of the masticatory muscles: subjects will be asked to hold their mandible in a resting position, without occlusal contact and avoiding swallowing, for ten seconds. The mean value will be considered the resting muscle activity, as described in the study by Martin et al.

Maximum voluntary contraction (MCV) in intercuspidation: subjects will be asked to clench their teeth as hard as possible for five seconds.

MCV in intercuspidation on cotton rolls: subjects will be asked to clench their teeth as hard as possible on cotton rolls positioned from the mandibular first molar to the mandibular canine on both sides, for five seconds.

From these last two tests (b and c), the samples with the highest root mean square (RMS) value will be used to calculate the indices. The electromyographic waveforms of each muscle with and without cotton rolls will be superimposed sample by sample, and the ratio between the superimposed areas and the total areas will be automatically calculated via software. This protocol was described by Ferrario et al. Therefore, for each subject, the sEMG potentials collected during MCV will be expressed as a percentage of the mean RMS potential collected during MCV on cotton rolls.

The dynamic tests will be as follows:

Chewing gum on the left side for fifteen seconds. Chewing gum on the right side for fifteen seconds.

To prevent the results from being affected by fatigue, a rest period of at least two minutes shall be allowed between static and dynamic tests.

Rapid Maxillary Expansion:

Subjects in the experimental group (with unilateral posterior crossbite) will be treated with Maxillary Rapid Expansion using a disjunctor fixed with two bands on the upper first permanent molars and a mesh cemented to the upper first premolars or upper first primary molars (depending on the eruptive stage of the patient). All the disjunctors will be manufactured and supplied by the same prosthetic laboratory (Corus Mondental, Castellar del Vallès, Barcelona). The bands will be fixed with glass ionomer cement (Ketac Cem Easymix; 3M ESPE, Saint Paul, Minnessotta, USA). The mesh will be cemented by preparing the enamel with 37% orthophosphoric acid (Octacid; Laboratorios Clarben S.A., Madrid, Spain), using a light-curing adhesive after washing and drying (Transbond XT; 3M Unitek, Saint Paul, Minnessotta, USA) and a light-curing flowable resin (Tetric EvoFlow; Ivoclar Vivadent AG, Schaan, Liechtenstein).

The breaker screw will be activated twice in the dental chair (0.5 mm). The patient's guardian will be trained to give two activations of the screw per day (0.5 mm). During the active disjunction phase, patients will be monitored once a week. The screw will be activated twice a day until a transverse overcorrection of 2 mm is achieved in the first permanent molars. When the active disjunction phase is completed, the screw will be blocked out with light-curing flowable resin (Tetric EvoFlow; Ivoclar Vivadent AG, Schaan, Liechtenstein) and the patient will wear the cemented disjunctor as a retainer for a minimum of six months.

The surface electromyographic activity (sEMG) of the anterior masseter and temporalis muscles will be recorded by means of the static and dynamic tests previously explained, before starting treatment (T0) in both the control and experimental groups. In the experimental group, the sEMG will also be recorded once the MCPU is already corrected with the disjunctor still cemented in the mouth (T1) and six months later, when the retention phase ends and the disjunctor is removed (T2).

ELIGIBILITY:
Inclusion Criteria:

* Mixed or early permanent dentition.
* Complete eruption of the first four permanent molars.
* Angle Class I ±1 mm.

Exclusion Criteria:

* Systemic diseases or congenital anomalies affecting craniofacial growth or development.
* Signs or symptoms of temporomandibular disorder (TMD).
* Dental pain.
* Previous orthodontic treatment.

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Muscle activity (microVolts) | change between baseline and 1 week follow-up; change between baseline and 6 months follow-up.
  sEMG is a NON-invasive method that measures the electrical activity of the muscle generated by the passage of the nerve impulse, which causes depolarization of the muscle cell membrane during excitation. Once the muscle is contracted and receives electrical signals, the electrodes pick up these signals and record them on the device application.
percentage of overlapping coefficient (%) | change between baseline and 1 week follow-up; change between baseline and 6 months follow-up.
  The standardized EMG waves of the left and right anterior temporalis (AT) and masseters (MM) were compared by computing a percentage overlapping coefficient (POC, unit: %, range: 0-100 per cent, norm values 85 per cent ≤ POC ≤ 100 per cent). If the muscles contract with perfect symmetry, a POC of 100 per cent (perfect symmetry) is expected. Conversely, a value corresponding to 0 per cent indicates the absence of concurrent activation of paired muscles (no symmetry). Three indices were computed for each subject (POC AT, POC MM and POC medium).
torque coefficient | change between baseline and 1 week follow-up; change between baseline and 6 months follow-up.
  This index is obtained by measuring the overlapping activity (standardized EMG waves) between the left MM and right AT and the right MM and left AT. The higher muscular activity of one couple (i.e. left MM and right AT) over the other (i.e. right MM and left AT) results in a torquing effect on the lower jaw. TC ranges between 0 per cent (no symmetric activation of the couples, greatest torquing effect) and 100 per cent (perfect symmetric activation of the couples, no torquing effect). Normal values are 90 per cent ≤ TC ≤ 100 per cent.
Total standardized muscle activity | change between baseline and 1 week follow-up; change between baseline and 6 months follow-up.
  This index is computed as the integrated area of the EMG standardized potentials of both MM and AT over time (5 seconds MVC). Norm values are 85 per cent ≤ IC ≤ 115 per cent. Lower values indicate that the EMG standardized potentials were reduced during the clenching tasks, and that the maximal EMG activity could not be expressed
Asymmetry index | change between baseline and 1 week follow-up; change between baseline and 6 months follow-up.
  This index is calculated by comparing the activity of the right couple (right AT and right MM) to the left couple (left AT and left MM). ASIM ranges from -100 per cent and +100 per cent; a value of 0 per cent depicts a perfect symmetric activation of the two couples. A negative value indicates greater activity of the left couple; conversely, a positive value indicates a greater activity of the right couple. Norm values are -10 per cent ≤ ASIM ≤ +10 per cent.
Symmetrical mastication index | change between baseline and 1 week follow-up; change between baseline and 6 months follow-up.
  assess whether the left and the right side chewing tests were performed with symmetrical muscular patterns. It indicates the distance between the centre of the chart and the centre of the ellipse in a graph that describes the prevalence of one side over the other during mastication. SMI ranges between 0 per cent (no symmetry) and 100 per cent (symmetrical muscular pattern). Normal values are 70 per cent ≤ SMI ≤ 100 per cent.
side of prevalent mastication | change between baseline and 1 week follow-up; change between baseline and 6 months follow-up.
  in case of SMI values lower than 70 per cent, the dominant side of mastication was identified as side of prevalent mastication. Three categories could be identified, that is right, left and symmetric.
frequency index | change between baseline and 1 week follow-up; change between baseline and 6 months follow-up.
  measures the frequency of masticatory cycles during the chewing experimental tasks and was reported in hertz (Hz: bites per second)

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional Catalunya, Barcelona, Sant Cugat, Spain